CLINICAL TRIAL: NCT00330616
Title: Clinical Evaluation of Bupropion SR (323U66)in Patients With Depression - Investigation in Elderly Patients With Depression
Brief Title: Study Of Bupropion SR (323U66) In Patients With Major Depressive Disorder In Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Masking: None | Purpose: Treatment
Other Study IDs: AK1102369
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2009-03-20 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2009-06

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: WELLBUTRIN; elderly; depression; Pharmacokinetics
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Drug: 323U66 SR

SUMMARY:
This is a study to obtain clinical experience of 323U66 SR for elderly patients with depression in repeat-dose of 323U66 SR up to 300mg/day, and to conduct exploratory investigation on safety, efficacy and pharmacokinetics profile in elderly patients with depression.

ELIGIBILITY:
Inclusion criteria:

* Target disease: Patients diagnosed as having the following primary disease and current major depressive episode for at least 8 weeks on the basis of DSM-IV-TR criteria.

  * Major Depressive Disorder, Single Episode (296.2x) (excluding those with psychotic features)
  * Major Depressive Disorder, Recurrent (296.3x). (excluding those with psychotic features)
* HAM-D (17 items) total score >/=18.
* Age: >/=65 years old (at the time of informed consent)
* Gender: Male or female.
* Inpatient or outpatient status: Either
* Informed consent: The subject himself/herself must give written informed consent.

Exclusion criteria:

* Patients with predisposition to seizure (who currently have or have a past history of seizure, febrile convulsive seizure in infancy, cerebral tumour, cerebrovascular disorder or head injury, who have a family history of idiopathic seizure, patients with diabetes who have been treated with oral hypoglycaemics or insulin, or who use drugs lowering the threshold of seizure)
* Patients who currently have or have a past history of the following disorders:

  * Anorexia nervosa (DSM-IV-TR 307.1)
  * Bulimia nervosa (DSM-IV-TR 307.51)
* Patients with a history of manic episode
* Patients with a past or current DSM- IV-TR diagnosis of schizophrenia or other psychotic disorder
* Patients with a current DSM-IV-TR Axis II diagnosis (e.g., antisocial or borderline personality disorder)
* Patients starting psychotherapy (except for supportive psychotherapy not aimed at therapeutic efficacy and unlikely to affect efficacy evaluation) and standardized cognitive behaviour therapy within 12 weeks prior to the start of the treatment phase
* Patients with a diagnosis of substance abuse (alcohol or drug) by the DSM-IV-TR criteria or with a diagnosis of substance dependence within 1 year prior to the start of the treatment phase
* Patients who have received electroconvulsive therapy within 24 weeks prior to the start of the treatment phase
* Patients who have taken MAO inhibitors (selegiline hydrochloride) within 2 weeks prior to the start of the treatment phase
* Patients who have taken another investigational drug within 12 weeks prior to the start of the pre-treatment phase
* Patients who have attempted suicide within 24 weeks prior to the start of the treatment phase, or patients for whom the score of the suicide-related item of HAM-D is >/=3, or patients in whom the risk of suicide is judged to be high by the investigator (sub-investigator).
* Patients in whom the risk of homicide is judged to be high by the investigator (sub-investigator).
* Patients with a history of hypersensitivity to 323U66
* Patients with serious cerebral disease
* Patients who have ECG or clinical evidence of any cardiac condition that the investigator (sub-investigator) assesses the subject is predisposed to ischemia or arrhythmia
* Patients with serious physical symptoms (i.e. cardiac/hepatic/renal disorder, hematopoietic disorder).

The index of seriousness is Grade 3 of "Criteria for classification of seriousness of adverse drug reactions to pharmaceutical products, etc." (PAB/PSD No.80 in 1992).

* Patients who have a history or complicated carcinoma or malignant tumour.
* Patients whose major depressive disorder is due to direct physiological effects of a general medical condition (for example, hypothyroidism, Parkinson's disease, chronic pain)
* Patients with systolic blood pressure of >/=160 mmHg or diastolic blood pressure of >/=100 mmHg at the start of the Treatment Period
* Patients diagnosed with dementia
* Patients who are inappropriate for participating in the study in the judgement of the investigator (sub-investigator).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion SR: Dose level 1 = 100mg tablet of Bupropion SR morning, after one week dose 1, increased to Dose 2 twice daily 100mg of Bupropion SR morning and evening, after one week at dose 2 could increase to Dose 3 150mg Bupropion twice daily morning and evening. Subjects stayed at dose level 3 for 6 weeks if tolerated.
Period: Overall Study
Arm/Group | Bupropion SR
Started | 35
Completed | 14
Not Completed | 21
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bupropion SR
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Rating Scale for Depression (HAM-D) Total Score at Week 8
Description: The Hamilton Rating Scale for Depression (HAM D) contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM D score range from 0 (not ill) to 53 (severely ill).
Time Frame: Baseline and Week 8
Population: Full Analysis Set consisted of all subjects in the safety population who had baseline and at least on post-baseline efficacy data and met the objectively-measured major eligibility criteria. Last observation carried forward method for missing data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 32
Scores on a scale | -8.4 (10.34)

2. Secondary Outcome: Percentage Change From Baseline in Hamilton Rating Scale for Depression (HAM-D) Total Score at Week 4
Description: The Hamilton Rating Scale for Depression (HAM D)contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM D score range from 0 (not ill) to 53 (severely ill).
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Bupropion SR
Number analyzed (Participants) | 17
Percentage of Change | -41.7 (25.40)

3. Secondary Outcome: Percentage Change From Baseline in Hamilton Rating Scale for Depression (HAM-D)Total Score at Week 8
Description: as for outcome 2
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Bupropion SR
Number analyzed (Participants) | 14
Percentage of Change | -60.7 (30.54)

4. Secondary Outcome: Percentage of Responders Based on the Hamilton Rating Scale for Depression (HAM-D) at Week 4
Description: The Hamilton Rating Scale for Depression (HAM D)contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM D score range from 0 (not ill) to 53 (severely ill). Responders are defined as subjects that had a decrease of >/= 50% total score on the HAM D.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Responders
Arm/Group | Bupropion SR
Number analyzed (Participants) | 17
Percentage of Responders | 29.4 (25.40)

5. Secondary Outcome: Percentage of Responders Based on the Hamilton Rating Scale for Depression (HAM-D) at Week 8
Description: as for outcome 4
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Responders
Arm/Group | Bupropion SR
Number analyzed (Participants) | 14
Percentage of Responders | 64.3

6. Secondary Outcome: Percentage of Remitters Based on the Hamilton Rating Scale for Depression (HAM-D) at Week 4
Description: The Hamilton Rating Scale for Depression (HAM D)contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM D score range from 0 (not ill) to 53 (severely ill). Remitters are defined as subjects with a HAM D total score of </= 7.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Remitters
Arm/Group | Bupropion SR
Number analyzed (Participants) | 17
Percentage of Remitters | 17.6 (30.54)

7. Secondary Outcome: Percentage of Remitters Based on the Hamilton Rating Scale for Depression (HAM-D) at Week 8
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Remitters
Arm/Group | Bupropion SR
Number analyzed (Participants) | 14
Percentage of Remitters | 50.0

8. Secondary Outcome: Change From Baseline in Hamilton Rating Scale for Depression (HAM-D) of Each Question's Score at Week 4
Description: as for outcome 2
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 17
Scores on a scale
  Depressed Mood | -1.4 (1.23)
  Feelings of Guilt | -0.7 (0.99)
  Suicide | -0.9 (1.03)
  Insomnia Early | -0.5 (0.87)
  Insomnia Middle | -0.5 (0.72)
  Insomnia Late | -0.6 (0.94)
  Work/Activities | -0.9 (1.17)
  Retardation | -1.2 (0.53)
  Anxiety Psychic | -0.9 (1.14)
  Anxiety Somatic | -0.8 (0.81)
  Somatic Symptoms GI | -0.3 (0.77)
  Somatic Symptoms General | -0.2 (0.90)
  Genital Symptoms | -0.5 (0.80)
  Hypochondriasis | -0.5 (0.94)
  Lose Weight History | -0.8 (0.88)
  Insight | -0.4 (0.62)

9. Secondary Outcome: Change From Baseline in Hamilton Rating Scale for Depression (HAM-D) for Each Question's Score at Week 8
Description: as for outcome 2
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 14
Scores on a scale
  Depressed Mood | -1.9 (1.46)
  Feelings of Guilt | -1.0 (1.11)
  Suicide | -1.1 (0.92)
  Insomnia Early | -0.9 (0.86)
  Insomnia Middle | -0.6 (0.74)
  Insomnia Late | -0.9 (0.86)
  Work/Activities | -1.4 (1.50)
  Retardation | -1.4 (0.63)
  Agitation | -0.5 (0.94)
  Anxiety Psychic | -1.5 (1.34)
  Anxiety Somatic | -1.1 (0.86)
  Somatic Symptoms GI | -0.6 (0.84)
  Somatic Symptoms General | -0.8 (0.89)
  Genital Symptoms | -0.6 (0.93)
  Hypochondriasis | -0.9 (1.07)
  Lose Weight History | -1.1 (1.21)
  Insight | -0.4 (0.63)

10. Secondary Outcome: Percentage of Change From Baseline in Hamilton Rating Scale for Depression (HAM-D)for Each Question's Score at Week 4
Description: The Hamilton Rating Scale for Depression (HAM-D)contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM-D score range from 0 (not ill) to 53 (severely ill).
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Bupropion SR
Number analyzed (Participants) | 17
Percentage of Change
  Depressed Mood | -47.1 (39.74)
  Feelings of Guilt | -76.7 (34.43)
  Suicide | -80.0 (36.84)
  Insomnia Early | -41.7 (59.67)
  Insomnia Middle | -40.6 (58.36)
  Insomnia Late | -42.9 (47.46)
  Work/Activities | -27.9 (31.86)
  Retardation | -73.5 (31.21)
  Agitation | -45.8 (68.28)
  Anxiety Psychic | -34.8 (43.72)
  Anxiety Somatic | -54.2 (39.67)
  Somatic Symptoms GI | -21.4 (57.89)
  Somatic Symptoms General | -17.9 (50.41)
  Genital Symptoms | -40.9 (62.52)
  Hypochondriasis | -38.1 (44.54)
  Lose Weight History | -57.7 (44.94)
  Insight | -60.0 (51.64)

11. Secondary Outcome: Percentage of Change From Baseline in Hamilton Rating Scale for Depression (HAM-D) for Each Question's Score at Week 8
Description: The Hamilton Rating Scale for Depression (HAM-D)contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM D score range from 0 (not ill) to 53 (severely ill).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Bupropion SR
Number analyzed (Participants) | 14
Percentage of Change
  Depressed Mood | -60.7 (40.62)
  Feelings of Guilt | -100.0 (0)
  Suicide | -83.3 (32.57)
  Insomnia Early | -70.0 (42.16)
  Insomnia Middle | -50.0 (61.24)
  Insomnia Late | -68.2 (46.22)
  Work/Activities | -42.3 (46.74)
  Retardation | -78.6 (32.31)
  Agitation | -52.8 (77.76)
  Anxiety Psychic | -55.4 (48.88)
  Anxiety Somatic | -60.7 (55.32)
  Somatic Symptoms GI | -45.8 (62.01)
  Somatic Symptoms General | -50.0 (60.30)
  Genital Symptoms | -45.5 (65.02)
  Hypochondriasis | -50.0 (43.23)
  Lose Weight History | -81.8 (33.71)
  Insight | -50.0 (70.71)

12. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D) Total Score at Week 4 and Week 8
Description: as for outcome 11
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 32
Scores on a scale
  Week 4 | 17.3 (6.94)
  Week 8 | 15.7 (8.41)

13. Secondary Outcome: Percentage of Responders Based on the Clinical Global Impression - Global Improvement Score (CGI-I)at Week 4 and Week 8
Description: The CGI-I assesses the investigator's impression of the patient's current illness. The time span is the week before the rating and the score ranges from 1 (very much improved) to 7 (very much worse). Responders are subjects that have a score of 1 (very much improved) or 2 (much improved) on the CGI-I.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Responders
Arm/Group | Bupropion SR
Number analyzed (Participants) | 33
Percentage of Responders
  Week 4 | 24.2
  Week 8 | 42.4

14. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity of Illness Score at Weeks 1, 2, 3, 4, 8
Description: The CGI-S assesses the investigator's impression of the severity of the patient's current illness. The time span is the week before the rating and the score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion SR
Number analyzed (Participants) | 34
Scores on a scale
  Week 1 | -0.2 (0.63)
  Week 2 | -0.4 (0.73)
  Week 3 | -0.4 (0.86)
  Week 4 | -0.6 (0.99)
  Week 8 | -0.9 (1.22)

15. Secondary Outcome: Adverse Events (>=5% Incidence)
Time Frame: Baseline through Week 8
Population: Safety population - all subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Bupropion SR
Number analyzed (Participants) | 35
Participants
  Nausea | 6
  Constipation | 5
  Dizziness | 5
  Nasopharyngitis | 4
  Pyrexia | 3
  Thirst | 3
  Weight Decreased | 3
  Glossitis | 2
  Paraesthesia Oral | 2
  Vomiting | 2
  Irritability | 2
  Oedema Peripheral | 2
  Somnolence | 2
  Blood Pressure Increased | 2
  Pruritus | 2
  Depression | 2
  Excoriation | 2
  Back Pain | 2

16. Secondary Outcome: Serious Adverse Events
Time Frame: Baseline through Week 8
Population: Safety population - all subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Bupropion SR
Number analyzed (Participants) | 35
Participants | 1

ADVERSE EVENTS:
Arm/Group | Bupropion SR
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 31
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Bupropion SR
Suicide attempt (Psychiatric disorders) | 1/35 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Bupropion SR
Nausea (Gastrointestinal disorders) | 6/35
Constipation (Gastrointestinal disorders) | 5/35
Dizziness (Nervous system disorders) | 5/35
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4/35
Pyrexia (General disorders) | 3/35
Thirst (General disorders) | 3/35
Weight decrease (Metabolism and nutrition disorders) | 3/35
Glossitis (Gastrointestinal disorders) | 2/35
Paraesthesia oral (Nervous system disorders) | 2/35
Vomiting (Gastrointestinal disorders) | 2/35
Irritability (Psychiatric disorders) | 2/35
Edema Peripheral (Blood and lymphatic system disorders) | 2/35
Somnolence (Psychiatric disorders) | 2/35
Blood Pressure increased (Cardiac disorders) | 2/35
Pruritus (General disorders) | 2/35
Depression (Psychiatric disorders) | 2/35
Excoriation (Skin and subcutaneous tissue disorders) | 2/35
Back Pain (General disorders) | 2/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.